CLINICAL TRIAL: NCT06486350
Title: Bone Marrow Supernatant IL-6 as a Predictor of Chemotherapy Sensitivity in AML Patients
Brief Title: IL-6: A Marker for AML Chemo Sensitivity
Status: Recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Huifang Huang, MD, Professor, Fujian Medical University Union Hospital
Other Study IDs: AML-IL6
Record Dates: First submitted 2024-06-19; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: AML, Adult
Keywords: AML; IL-6; Chemotherapy sensitivity
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bone marrow supernatant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute myeloid leukemia (AML) is a clonal malignancy that arises from the primitive hematopoietic cells within the hematopoietic system. According to SEER cancer statistics, the 5-year survival rate for AML patients stands at a concerning 30%. Despite therapeutic advancements, the development of chemotherapy resistance and the risk of disease relapse pose significant barriers to curative outcomes. Evidence has linked elevated interleukin-6 (IL-6) levels in plasma and bone marrow to a poorer prognosis in AML, with IL-6 potentially fostering chemotherapy resistance through the enhancement of fatty acid uptake and the induction of stromal-like morphological changes in AML cells. However, the role of IL-6 as a potential biomarker for monitoring chemotherapy sensitivity in AML has not been fully elucidated. This study seeks to investigate the correlation between IL-6 levels in bone marrow supernatant and the sensitivity to chemotherapy, offering a clinical perspective that could pave the way for improved prognostic markers and personalized treatment strategies.

DETAILED DESCRIPTION:
In this prospective study, we will collect bone marrow supernatant samples from patients diagnosed with Acute Myeloid Leukemia (AML) to evaluate the levels of Interleukin-6 (IL-6). Our aim is to explore whether elevated IL-6 levels can serve as a predictive biomarker for poor treatment outcomes following standard chemotherapy regimens. The findings may help in stratifying patient risk and personalizing therapeutic approaches in AML treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis aligns with the "Chinese guidelines for diagnosis and treatment of adult acute myeloid leukemia (not APL) (2023)";
2. All patients are experiencing their first onset of the disease and have not received any related chemotherapy prior to the study;
3. Patients participate in the study accompanied by family members and sign informed consent documents.

Exclusion Criteria:

1. Patients with concurrent malignancies requiring treatment;
2. Presence of infectious diseases, including SARS, viral hepatitis, or HIV/AIDS;
3. Major surgery performed within the last 21 days;
4. Performance Status (PS) score >3;
5. Severe liver or kidney dysfunction or serious infection;
6. Severe psychiatric conditions that impair understanding of the study protocol or voluntary withdrawal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective study enrolls patients who fulfill the diagnostic criteria for AML (excluding APL), with an age requirement of over 18 years and no restrictions on gender. Participation is entirely voluntary, with each participant or their legal guardian being thoroughly informed about the study details and signing an informed consent form. Participants are willing to adhere to and capable of completing all required study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  The primary endpoint of this study is the overall response rate (ORR) after Chemotherapy

SECONDARY OUTCOMES:
CR | 1 year
  The secondary endpoints is the complete remission (CR) rate after Chemotherapy
CRi | 1 year
  The secondary endpoints is the complete remission with incomplete blood count recovery (CRi) rate after Chemotherapy
PR | 1 year
  The secondary endpoints is the partial remission (PR) rate after Chemotherapy
OS | 2 year
  The secondary endpoints is the overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hou D, Cai D, Dai W, Liao X, Tan M, Zheng X, Wang L, Liu J, Wang J, Wang X, Fu Q, Huang H. Targeting bone marrow mesenchymal stromal cell-derived IL-6 to overcome acute myeloid leukemia chemoresistance. Blood Adv. 2025 Oct 14;9(19):4810-4824. doi: 10.1182/bloodadvances.2024015496. PMID 40668612